CLINICAL TRIAL: NCT02431065
Title: Comparing the Analgesic Effects of Ultrasonography-guided and Direct-surgical Rectus Sheath Block in Single-port Access Laparoscopy Patients
Brief Title: Ultrasonography-guided and Surgical Rectus Sheath Block in Single-port Access Laparoscopy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chungnam National University Hospital (Other)
Responsible Party: Principal Investigator, Heon-Jong Yoo, Clinical Vice professor, Chungnam National University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GyAne-1
Record Dates: First submitted 2015-04-17; First posted 2015-04-30 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Pain
Keywords: Rectus sheath block; Single port laparoscopy
MeSH Terms: conditions — Pain | interventions — Anesthesia; Ropivacaine; Surgical Procedures, Operative; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 3, Direct injection group (Experimental): Test group 2, Rectus sheath block will be performed under direct visualization. Ropivacaine (0.75%, 10ml) will be directly injected into the right and left rectus sheath at the end of the operation.
  Interventions: Procedure: Rectus sheath block; Drug: Ropivacaine
- Group 2, ultrasonography group (Active Comparator): Test group 1, Rectus sheath block will be performed under sonographic guidance. Ropivacaine (0.75%, 10ml) will be injected into the right and left rectus sheath under ultrasonographic guidance at the end of the operation.
  Interventions: Procedure: Rectus sheath block; Drug: Ropivacaine
- Group 1 (Placebo Comparator): Control group, Rectus sheath block will be performed under sonographic guidance. Normal saline 10 ml will be injected into the right, left rectus sheath under ultrasonography guidance at the end of the operation.
  Interventions: Procedure: Rectus sheath block; Other: Normal saline

INTERVENTIONS:
Procedure: Rectus sheath block — Local anesthetics (Ropivacaine 0.75% 10ml) or normal saline (10ml) will be injected in the rectus sheath via different methods:
  1. Control group Normal saline 10mL will be injected under ultrasonography guidance into the right, left rectus sheath at the end of the operation before emergence from general anesthesia.
  2. Ultrasonography group Local anesthetic (Ropivacaine 0.75% 10 mL) will be injected under ultrasonography guidance into the right left rectus sheath at the end of the operation before emergence from general anesthesia.
  3. Direct injection group Local anesthetic (Ropivacaine 0.75% 10 mL) will be injected under direct visualization into the right, left rectus sheath at the end of the operation before emergence from general anesthesia.
  Other Names: anesthesia
Drug: Ropivacaine — Local anesthetics (Ropivacaine 0.75% 10ml) or normal saline (10ml) will be injected in the rectus sheath via different methods:
  1. Control group Normal saline 10mL will be injected under ultrasonography guidance into the right, left rectus sheath at the end of the operation before emergence from general anesthesia.
  2. Ultrasonography group Local anesthetic (Ropivacaine 0.75% 10 mL) will be injected under ultrasonography guidance into the right left rectus sheath at the end of the operation before emergence from general anesthesia.
  3. Direct injection group Local anesthetic (Ropivacaine 0.75% 10 mL) will be injected under direct visualization into the right, left rectus sheath at the end of the operation before emergence from general anesthesia.
  Other Names: surgery
  Arms: Group 2, ultrasonography group; Group 3, Direct injection group
Other: Normal saline — Local anesthetics (Ropivacaine 0.75% 10ml) or normal saline (10ml) will be injected in the rectus sheath via different methods:
  1. Control group Normal saline 10mL will be injected under ultrasonography guidance into the right, left rectus sheath at the end of the operation before emergence from general anesthesia.
  2. Ultrasonography group Local anesthetic (Ropivacaine 0.75% 10 mL) will be injected under ultrasonography guidance into the right left rectus sheath at the end of the operation before emergence from general anesthesia.
  3. Direct injection group Local anesthetic (Ropivacaine 0.75% 10 mL) will be injected under direct visualization into the right, left rectus sheath at the end of the operation before emergence from general anesthesia.
  Other Names: No intervention
  Arms: Group 1

SUMMARY:
Rectus sheath block is effective in reducing pain in the peri-umbilical region, and the use of ultrasonography is recommended to perform the block at the precise location. Recently, intra-operative rectus sheath block has also been introduced without the aid of ultrasonography. However, no study has not yet compared the analgesic effects of these two different approaches (ultrasonography-guided vs direct surgical). Thus, the aim of our study is to compare the effect of ultrasonography-guided and direct-surgical rectus sheath block after single-port access laparoscopy in benign ovary cyst patients.

DETAILED DESCRIPTION:
This is a randomized, prospective study comparing the analgesic effects of ultrasonography-guided and direct-surgical rectus sheath block after single-port access laparoscopy in benign ovary cyst patients.

Patients will be randomly divided into 3 groups based on the procedure: control group, ultrasonography group and direct injection group. Each group consists of 30 patients.

* Control group Normal saline 10mL will be injected under ultrasonography guidance into the right, left rectus sheath at the end of the operation before emergence from general anesthesia.

  * Ultrasonography group Local anesthetic (Ropivacaine 0.75% 10 mL) will be injected under ultrasonography guidance into the right left rectus sheath at the end of the operation before emergence from general anesthesia.

    * Direct injection group Local anesthetic (Ropivacaine 0.75% 10 mL) will be injected under direct visualization into the right, left rectus sheath at the end of the operation before emergence from general anesthesia.

Analgesic efficiency will be assessed using the VAS (visual analogue scale) pain scale and the total amount of self-administered fentanyl via PCA (patient controlled analgesia) devices at multiple time scales (1, 6, 10, 24 and 48 hours after surgery). We will also compare the incidence of fentanyl complications, such as nausea, vomiting, pruritus and dizziness

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for a single port laparoscopic surgery at Chung Nam University hospital due to benign tumor of the ovary or the fallopian tube
2. Between age of twenty to seventy
3. Patients with a physical rating of 1 or 2 according to the American Anesthesiology guidelines
4. Patients who have not had laparoscopic surgery within two months

Exclusion Criteria:

1. Hysterectomy via single port laparoscopic surgery
2. Patients with chronic pelvic pain
3. Abdominal pain of unknown origin
4. Suspected malignant tumor
5. Diagnosed with malignant tumor of any origin
6. Patients currently taking psychiatric medicine
7. Pregnancy
8. Patients with a history of hypersensitivity to amide type local anesthetics
9. Patients with a history of hypersensitivity to opioid
10. Risk of bleeding
11. Unable to comprehend or does not agree to the consent form

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
The intensity of pain as assessed by Dose of fentanyl(opioid) | within 24 hours of surgery
  Dose of fentanyl(opioid) self-administered by the patients within 24 hours of surgery

SECONDARY OUTCOMES:
Incident rate of side effects of fentanyl | within 24 hours of surgery
  Incident rate of side effects of fentanyl including nausea and vomiting by the patients within 24 hours of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Heon Jong Yoo, MD. PhD, Principal Investigator — Chung Nam National University Hospital, clinical vice professor

REFERENCES:
- [Background] Crosbie EJ, Massiah NS, Achiampong JY, Dolling S, Slade RJ. The surgical rectus sheath block for post-operative analgesia: a modern approach to an established technique. Eur J Obstet Gynecol Reprod Biol. 2012 Feb;160(2):196-200. doi: 10.1016/j.ejogrb.2011.10.015. Epub 2011 Nov 21. PMID 22104479
- [Background] Osaka Y, Kashiwagi M, Nagatsuka Y, Oosaku M, Hirose C. [Ultrasound-guided rectus sheath block for upper abdominal surgery]. Masui. 2010 Aug;59(8):1039-41. Japanese. PMID 20715537